CLINICAL TRIAL: NCT05619913
Title: The EPOCH Study: Phase II Open Labelled Study Investigating the Use of Single Agent Eribulin and Eribulin in Combination With Pembrolizumab in Relapsed Tubo-ovarian or Uterine Carcinosarcoma
Brief Title: EPOCH: Eribulin and Pembrolizumab in Ovarian/Uterine Carcinosarcoma
Acronym: EPOCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australia New Zealand Gynaecological Oncology Group (Other)
Collaborators: Eisai Inc. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZGOG 1828/2021
Record Dates: First submitted 2022-10-26; First posted 2022-11-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Carcinosarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — eribulin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - Single agent eribulin arm (Experimental): Eribulin until progression of disease (PD) as defined by RECIST v1.1, unacceptable toxicity or physician/patient discretion or choice to cease treatment.
  Patients who progress on the single agent eribulin arm may receive combination eribulin and pembrolizumab.
  Interventions: Drug: Eribulin Mesylate
- Arm 2 - Combination eribulin and pembrolizumab arm (Experimental): Eribulin for a maximum of 6 cycles. Pembrolizumab until PD or a maximum of 35 cycles (including the 6 cycles where it is administered in combination with eribulin) or until unacceptable toxicity or physician/patient discretion or choice to cease treatment.
  Interventions: Drug: Eribulin Mesylate; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesilate is a first-in-class halichondrin B-based, microtubule dynamics inhibitor7. It inhibits the growth phase of microtubules without affecting the shortening phase and sequesters tubulin into non-productive aggregates.
  Other Names: Halaven
Drug: Pembrolizumab — Pembrolizumab is a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD 1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2).
  Other Names: Keytruda
  Arms: Arm 2 - Combination eribulin and pembrolizumab arm

SUMMARY:
The EPOCH study population is patients with tubo-ovarian carcinosarcoma or uterine carcinosarcoma with evidence of recurrence or progression.

The study aims to determine the activity of eribulin as a single agent and the combination of eribulin and pembrolizumab as measured by clinical benefit rate (CBR) at 12 weeks.

Additionally, the study aims to establish whether high mobility group A2 (HMGA2) protein expression is a good functional biomarker to predict response to eribulin and pembrolizumab.

DETAILED DESCRIPTION:
EPOCH (Eribulin and Pembrolizumab in Tubo-Ovarian and Uterine Carcinosarcoma) is an international clinical trial, which aims to improve outcomes in people with the rare and highly lethal Ovarian Carcinosarcoma (OCS) or Uterine Carcinosarcoma (UCS) malignancies.

The underlying study rationale is based on robust preclinical evidence that demonstrated that eribulin, a microtubule inhibitor, can reprogram the tumour microenvironment, reversing epithelial mesenchymal transition (EMT) in these mesenchymal cancers, and potentiate the response to immune checkpoint blockade.

In addition, expression of HMGA2, a high mobility group protein has been associated with activation of EMT process and may be a predictive biomarker of eribulin-responsive cancers. This study is aimed at translating these laboratory findings to the clinic and treat patients with recurrent OCS and UCS with eribulin and the immune checkpoint inhibitor pembrolizumab, which targets and blocks the programmed cell death receptor 1 (PD-1).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures and the ability to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations.
2. Patients > 18 years old who have a histologically confirmed tubo-ovarian carcinosarcoma or uterine carcinosarcoma with evidence of recurrence or progression. The component of sarcoma in the diagnostic pathology sample must be equal to or > 5% of tumour.
3. Must have Positron Emission Tomography (PET), Computerized Tomography CT, or Magnetic Resonance Imaging (MRI) -proven relapsed disease after completion of at least one line and not more than two lines of chemotherapy.
4. Must have at least one evaluable measurable lesion (other than the lesion that will be used for biopsy) using standard techniques according to the Response Evaluation Criteria in Solid Tumours (RECIST v1.1) guidelines (Appendix 1).
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (Appendix 5). Evaluation of ECOG is to be performed within 28 days prior to the first dose of the study intervention.
6. Have adequate organ function as defined below (refer also Appendix 6).

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelets ≥100 x 109/L
   * Haemoglobin (Hb) ≥90 g/L or ≥5.6 mmol/L (criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks).
   * Creatinine ≤ 1.5 x Upper Limit Normal (ULN); OR Creatinine Clearance (CrCl) ≥ 30 mL/min (calculated per institutional standard) for participants with creatinine levels >1.5 ULN (glomerular filtration rate, GFR, can also be used in place of creatinine or CrCl). (Patients with moderate renal impairment (CrCl 30-49ml/min) will receive a 25% reduced dose of eribulin).
   * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
   * Alkaline phosphatase (ALP), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
   * International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants Biological specimens must be collected within 28 days prior to the first dose of the study intervention (within 7 days, where indicated in the SoA).
7. Available formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer and/or metastatic tumour from the up-front or secondary debulking surgery with adequate neoplastic cell content (>30%).
8. Must have disease amenable to biopsy and must be willing to undergo a paired biopsy for additional correlative analyses (the first biopsy to be performed within 28 days prior to the start of the study intervention and the second biopsy in the five-day window prior to Cycle 2 (post Cycle 1)). For patients that experience progression of their disease whilst on study, separate patient consent will be sought for additional biopsies of their tumour for research.
9. Willing to have blood samples collected for translational research
10. Must not be pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a person of childbearing potential (POCBP). OR
    2. A POCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 months (120 days) after the last dose of the study treatment.

Exclusion Criteria:

1. Prior line of treatment involving immunotherapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor. This criteria is applicable for both intervention arms as patients may cross-over from the non-immunotherapy arm during their study participation.
2. Prior treatment with eribulin for any malignancy.
3. Absence of a second disease site suitable for biopsy
4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the first dose of the study intervention.
5. Has active autoimmune disease (such as Systemic Lupus Erythematosus) that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
6. A POCBP who has a positive urine pregnancy test within 7 days prior to the first dose of the study intervention (see Appendix 7). If the urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Has received prior radiotherapy within 2 weeks of the start of the study intervention. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease.
8. Known central nervous system malignancy or metastasis, including leptomeningeal metastasis or carcinomatous meningitis, unless adequately treated and patients are neurologically stable for at least one month prior to enrolment. Patients must be either off corticosteroids or on stable or decreasing dose of < /=10 mg daily prednisone (or equivalent) within 28 days prior to the first dose of the study intervention. In the case of short-term use of systemic corticosteroids (less than 24 hours within 28 days) of greater than 10 mg daily of prednisone or an equivalent corticosteroid, the required washout period prior to starting the first dose of the study intervention is 7 days. Anticonvulsants are allowed to be continued except for those which interfere with the study interventions or are associated with liver toxicity. However, patients receiving anticonvulsants must be discussed with Study Chair or Acting Chair of Trial Management Committee (TMC) prior to their enrolment to the study.
9. Symptomatic or clinically significant inflammatory bowel disease (Crohn's disease or ulcerative colitis).
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study intervention.
11. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of the study intervention. Live vaccine or live-attenuated vaccine cannot be administered during treatment with the study intervention and for 30 days post discontinuation of the study intervention. Administration of killed vaccines is allowed.
12. Has an active infection requiring systemic therapy.
13. Has had an allogenic tissue/solid organ transplant.
14. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
15. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
16. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: no testing for HIV is required unless mandated by local health authority.
17. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA > 25 international units/mL is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
18. Has a known additional active malignancy that is likely to interfere with assessment of response or tolerance to the study intervention.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patients' participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
20. Inability to attend or comply with treatment or follow-up scheduling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) by RECIST v1.1 in combination therapy arm | 12 Weeks
  CBR defined as Partial Response (PR), Complete Response (CR) or Stable Disease (SD) by RECIST v1.1 in the combination therapy arm.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 in single agent therapy arm | 12 weeks
  CBR defined as Partial Response, Complete Response or Stable Disease by RECIST v1.1 in the single agent therapy arm.
Objective Response Rate (ORR) in both the single agent eribulin and combination eribulin/pembrolizumab arms | 12 weeks
  Objective Response Rate (CR and PR by RECIST v1.1) at 12 weeks in both the single agent eribulin and combination eribulin/pembrolizumab arms
Clinical Benefit Rate (CBR) by iRECIST (modified RECIST guidelines for use in cancer immunotherapy trials) | 12 weeks
  Clinical Benefit Rate (CR and PR and SD) by irRECIST at 12 weeks in both the single agent eribulin and combination eribulin/pembrolizumab arms
Time to progression in the combination therapy arm | Up to 3 years
  Determine time to progression in the combination therapy arm
Progression free survival (PFS) | Up to 4 years
  Determine progression free survival (PFS)
Overall Survival (OS) | Up to 4 years
  Determine Overall Survival (OS)
Adverse events | Up to 4 years
  Determine toxicity, frequency, and severity of Adverse Events (CTCAE V5.0)
Health related Quality of Life using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for cancer patients (QLQ C30) | Up to 4 years
  Determine aspects of health-related quality of life using EORTC QLQ C30
Health related Quality of Life using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire module for Ovarian Cancer patients (OV28) | Up to 4 years
  Determine aspects of health-related quality of life using EORTC OV28

OTHER OUTCOMES:
Duration of response | Up to 4 years
  Duration of response represented in annotated swimmers plot
High mobility group A2 (HMGA2) protein expression | Up to 4 years
  Evaluate HMGA2 expression as predictive biomarker for response benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Scott, AM MB BS PhD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (6):
- Australia (4):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No